CLINICAL TRIAL: NCT00417573
Title: Efficacy of IgIv in Patients With IgG Subclass Deficiency and Recurrent Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Center for Rheumatic Disease, Allergy, & Immunology (Other)
Collaborators: Grifols Therapeutics LLC (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-489
Record Dates: First submitted 2006-12-28; First posted 2007-01-01 (Estimated); Last update posted 2007-01-01 (Estimated); Status verified 2006-12

CONDITIONS: IgG Deficiency; Infections
Keywords: Immunodeficiency; Gammaglobulin; IgG subclass deficiency with recurrent infections
MeSH Terms: conditions — IgG Deficiency; Infections; Immunologic Deficiency Syndromes

INTERVENTIONS:
Drug: IV Gamunex 10%

SUMMARY:
* This is the first study, that we are aware of, that will evaluate the efficacy of IgIV in patients with IgG subclass deficiency.
* Will provide data for further collaboration in extending study to involve other immunological centers in the United States to study patients with similar disease.

DETAILED DESCRIPTION:
*10 consenting adults (18 or older) will receive IgIV (Gamunex 10%) monthly at a dose of 400mg/kg body weight IV at 3ml/minute. Comprehensive labs will be monitored at each visit, as well as clinical eval, plus patients will complete a questionnaire each time. There is also a 3 month follow-up visit after completion of therapy. Specific xrays will be done at the beginning and with the last treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 or older) with deficiency in one or more IgG subclasses with documented history of recurrent infections limited to upper or lower respiratory tract, urinary, and/or skin.

Exclusion Criteria:

* Patients with panhypogammaglobulinemia or selective IgA deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2004-12; Study Completion 2006-12

PRIMARY OUTCOMES:
Lab values ck'ed baseline and with each treatment, and 15 mo. visit
Xray of Chest and sinus baseline and on 12th and last treatment
Clinical assessment baseline, every treatment, and 15 mo.

SECONDARY OUTCOMES:
Patient questionnaires completed by patients, baseline, prior to each treatment, and at 15 month vist.

CONTACTS AND LOCATIONS:
Overall Officials: Nabih I Abdou, MD, PhD, Principal Investigator — Center for Rheumatic Disease, Allergy, Immunology
Locations (1):
- Center for Rheumatic Disease, Allergy, Immunology, Kansas City, Missouri, United States

REFERENCES:
- [Derived] Abdou NI, Greenwell CA, Mehta R, Narra M, Hester JD, Halsey JF. Efficacy of intravenous gammaglobulin for immunoglobulin G subclass and/or antibody deficiency in adults. Int Arch Allergy Immunol. 2009;149(3):267-74. doi: 10.1159/000199723. Epub 2009 Feb 12. PMID 19218820